CLINICAL TRIAL: NCT00221780
Title: Importance of Left Ventricular Pacing Site in Biventricular Resynchronization Therapy for Severe Heart Failure
Brief Title: Role of Left Ventricular Pacing Site
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Ministry of Health, France (Other Government)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 9426-01; 2001-030
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2007-06-29 (Estimated); Status verified 2007-06

CONDITIONS: Heart Failure; Cardiomyopathy, Dilated; Coronary Disease
Keywords: Heart failure; Cardiomyopathy, dilated; Coronary disease; Cardiac Pacing, Artificial; Hemodynamics; Randomized Controlled Trials; Single-Blind Study
MeSH Terms: conditions — Heart Failure; Cardiomyopathy, Dilated; Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: left ventricular pacing

SUMMARY:
Cardiac resynchronization therapy has been shown to be effective in reducing symptoms and mortality in heart failure patients. However, very few is known about the importance of the left ventricular pacing site. We study in a random order 11 different left ventricular pacing sites and compare their hemodynamics using pressure-volume catheters. The consequences on the surface ECG are also assessed.

DETAILED DESCRIPTION:
Background. Cardiac resynchronization therapy has been shown to be effective in reducing symptoms and mortality in heart failure patients. However, very few is known about the importance of the left ventricular pacing site.

Design. Single-blind, monocentric, randomized cross-over study comparing 11 left ventricular pacing sites in a random order.

Intervention. Left ventricular DDD pacing on 11 ventricular sites, prior to the implantation. At each pacing site, a control hemodynamics will be obtained in AAI pacing at the same pacing rate. At each pacing site, 2 AV delays, a short and a long one, will be assessed.

Eligibility criteria. Patients referred for cardiac resynchronization therapy for heart failure

Outcomes. Hemodynamic measures using pressure-volume catheters.

ELIGIBILITY:
Inclusion Criteria:

* Heart failure referred for cardiac resynchronization therapy
* NYHA Class III or IV
* Informed consent form signed

Exclusion Criteria:

* Hypertension not controlled by treatment
* Coronary ischemia not controlled by treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2003-11; Study Completion 2007-12 (Estimated)

PRIMARY OUTCOMES:
Variation in left ventricular dp/dt max

SECONDARY OUTCOMES:
pressures and volumes of the left ventricle
stroke work
surface ECG repolarisation

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Jaïs, Dr, Principal Investigator — University Hospital, Bordeaux; Paul Perez, Dr, Study Chair — University Hospital, Bordeaux
Locations (1):
- Hôpital Cardiologique du Haut Lévêque, Rythmology department, Pr CLEMENTY, 3rd Floor, Pessac, France